CLINICAL TRIAL: NCT03785821
Title: Development and Clinical Application of Bitter Melon Seed Oil as a Functional Food for Treating Obesity and Hepatic Steatosis
Brief Title: Effect of Bitter Melon Seed Oil on Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CMUH104-REC3-014
Record Dates: First submitted 2018-12-13; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Weight Gain
Keywords: Bitter melon seed oil; Olive oil; Weight control; UCP1 polymorphism
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMSO (Experimental): Bitter melon seed oil supplementation
  Interventions: Dietary Supplement: BMSO
- OO (Placebo Comparator): Olive oil supplementation
  Interventions: Dietary Supplement: OO

INTERVENTIONS:
Dietary Supplement: BMSO — BMSO was extracted from Hualien No. 4 cultivate of bitter melon seed. BMSO were incorporated into capsules containing 0.5 g of oil. All persons took 3 capsules after each meal, i.e. 9 capsules (4.5 g of oil) daily, resulting in daily consumption of 2.3 g alpha-ESA in the BMSO group.
  Arms: BMSO
Dietary Supplement: OO — Olive oil (extra virgin grade) was purchased from La Espanola (Acesur, Spain). OO were incorporated into capsules containing 0.5 g of oil, identical appearance to BMSO. All persons took 3 capsules after each meal, i.e. 9 capsules (4.5 g of oil) daily.
  Arms: OO

SUMMARY:
To investigate the metabolic benefits of bitter melon seed oil (BMSO), overweight or obese healthy Taiwanese adults (n=60) were randomly assigned to receive capsules containing either olive oil (OO; placebo) or BMSO at 4.5 g/d dose for 12 week. Across intervention period, body weight, BMI, waist-to-hip ratio, and body fat mass were measured. Blood were collected before and after intervention for measurements of blood lipid and inflammatory cytokines. The anti-obesity effect of BMSO was further assessed by stratification of participants according to UCP1 rs1800592 polymorphism.

DETAILED DESCRIPTION:
Bitter melon is a common Asian vegetable. Its seed is not edible and discarded as a waste product. However, the seed oil is enriched in cis9, trans11, trans13-conjugated linolenic acid or alpha-eleostearic acid (alpha-ESA). Investigators previously demonstrated the anti-obesity functions of bitter melon seed oil (BMSO) in animal trials. Herein, a RCT was conducted to test the potential of BMSO in developing as a functional culinary oil for weight control.

Considering UCP-1 played a pivotal role in anti-adiposity function of BMSO as demonstrated in animal studies, the anti-obesity effect of BMSO was further assessed according to UCP1 rs1800592 polymorphism.

Healthy Taiwanese adults with overweight or obesity were recruited by advertisement and were assessed by a family medicine physician for eligibility. All participants signed the consent form. Blocked randomization was used to randomly assign participants into one of two groups to receive indicated supplement (BMSO or OO capsules with identical appearance; 4.5 g oil/d) for 12 week. Subjects were requested to maintain their usual diet and physical activity during the study period (0-12 week).

Anthropometric measurements were done on week 0, 4, 8 and 12. Three-day food records, collection of blood samples and physical health check were conducted on week 0, 4 and 12. Indirect calorimetry was done on week 0 and 12. Questionnaires about self-reported side effects, such as trouble sleeping, constipation, diarrhea, increased heartbeat, palpitations, headache, anxiety, or dizziness, were collected in each visit. Group allocation was concealed.

ELIGIBILITY:
Inclusion Criteria:

* adults with overweight or obesity (BMI ≥ 24 kg/m2 or waist circumference > 90 cm in males and > 80 cm in females)
* 20-64 y of age
* not currently using any weight-reducing agent

Exclusion Criteria:

* diabetes
* endocrine disease
* uncontrolled high blood pressure (systolic ≥ 180 mm Hg or diastolic ≥ 110 mm Hg)
* liver, kidney, or cardiovascular disease
* gastrointestinal disease
* psychological diseases
* pregnancy or lactation
* asthma and allergies
* smoking
* use of any drugs or dietary supplements that potentially affected body weight, blood lipids, blood pressure, or inflammatory responses.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Weight gain | 12 week
  Changes at intervention for 4,8 and 12 week

SECONDARY OUTCOMES:
BMI | 12 wk
  Changes at intervention for 4,8 and 12 week
waist-to hip ratio | 12 wk
  Changes at intervention for 4,8 and 12 week
body fat mass | 12 wk
  Changes at intervention for 4,8 and 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Min Chao, PhD, Principal Investigator — China Medical University, China

IPD SHARING:
Plan to Share IPD: No